CLINICAL TRIAL: NCT04740294
Title: Efficacy of Magnesium Sulfate Bolus in Pediatric Patients With Bronchiolitis
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, John W Berkenbosch, Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20.1171
Record Dates: First submitted 2021-02-01; First posted 2021-02-05 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Bronchiolitis, Viral
MeSH Terms: conditions — Bronchiolitis, Viral | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This is a randomized placebo-controlled pilot study with 1:1 randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be done in the pharmacy using a pre-developed randomization table. Study medication, whether MgSO4 or placebo, will be prepared by a study pharmacist and sent to the nursing/clinical staff for administration labelled as "study drug". Unblinding, if clinically indicated, can be provided to the treatment team but it is not anticipated that this will be required.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Magnesium Sulfate (Experimental): The patient will receive a bolus of 50mg/kg MgSO4 over twenty minutes.
  Interventions: Drug: Magnesium Sulfate
- Placebo (Placebo Comparator): The patient will receive a bolus of Normal Saline over twenty minutes.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Randomized to receive either magnesium sulfate or normal saline placebo.

SUMMARY:
The purpose of this study is to more rigorously evaluate the response to a single bolus of magnesium sulfate in a population of patients with moderate to severe bronchiolitis. The primary outcome will be to evaluate the effect of this therapy on clinical respiratory status. Secondary outcomes of interest will include the incidence of adverse effects and safety profile of magnesium bolus use in this population.

DETAILED DESCRIPTION:
This randomized placebo-controlled pilot study is designed to evaluate the above referenced outcomes. Study drug initiation will occur in the local pediatric intensive care unit in patients with a clinical diagnosis of bronchiolitis and whose parent/LAR consents for their participation. Our goal is to enroll and evaluate a total of 40 patients.

Upon obtaining informed consent, the participant will receive an enrollment history and physical to include: baseline Modified Pulmonary Index Score (MPIS), blood pressure, vital signs, and epidemiologic data. The participant will then receive either a bolus of 50mg/kg Magnesium Sulfate (MgSO4) or normal saline as placebo medication over twenty minutes. Vital signs and MPIS will be monitored according to the study schedule, for a total of six hours. During the period of monitoring subjects will not receive additional bronchodilators unless otherwise deemed clinically necessary by the subject's attending physician. If administered, these will be recorded by investigative team.

ELIGIBILITY:
Inclusion Criteria:

* Infants under 12 months of age
* Admitted to the pediatric intensive care unit
* Moderate/severe bronchiolitis using MPIS
* Less than 24 hours of admission to the PICU
* Parent/LAR consents for infant to participate

Exclusion Criteria:

* Patients with the following conditions are ineligible: chronic lung disease, unrepaired congenital heart disease, and cyanotic heart disease.

Ages: 1 Month to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-07-21 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of this therapy on clinical respiratory status | 6 hours post bolus of medication versus placebo
  MPIS will be used to follow respiratory status

SECONDARY OUTCOMES:
Identify the incidence of adverse effects and safety profile of magnesium sulfate | 6 hours post bolus of medication versus placebo
  Patients will be followed for any potential adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: John W Berkenbosch, MD, Principal Investigator — University of Louisville
Locations (1):
- Norton Children's Hospital, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
The information will not be shared outside of the University except as de-identified data for presentation of results virtually or in print.